CLINICAL TRIAL: NCT00372684
Title: PALUREA: Severe Falciparum Imported Malaria in Adults: Clinical and Physiopathological Study
Brief Title: PALUREA: Severe Imported Malaria in Adults
Acronym: PALUREA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Christophe AUCAN, Department Clinical Research of developpement
Other Study IDs: P051063; AOR05007
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2007-07

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Malaria; Imported malaria; Severe malaria; Uncomplicated malaria; Intensive Care Units; Polymorphism, Genetic; Parasitic Sensitivity Tests; Inflammation Mediators
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Intensive Care Units

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — physiopathologic
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: with severe malaria hospitalized in ICU
  Interventions: Genetic: with severe malaria hospitalized in ICU
- 2: with uncomplicated malaria
  Interventions: Genetic: with uncomplicated malaria

INTERVENTIONS:
Genetic: with severe malaria hospitalized in ICU — with severe malaria hospitalized in ICU
  Groups: 1
Genetic: with uncomplicated malaria — with uncomplicated malaria
  Groups: 2

SUMMARY:
Plasmodium falciparum malaria remains a major public health problem in endemic areas, with approximately 2 million deaths each year, especially in tropical African countries.

In non-endemic industrialized areas, imported malaria is generally diagnosed in travelers, as well as immigrants from endemic countries. Such imported cases have increased worldwide, with approximately 7000 cases each year in France. Among these cases, 300 are severe requiring hospitalization in the intensive care unit (ICU) with an overall mortality rate of 10%, despite available effective care.

Many studies have been performed to evaluate clinical and physiopathological aspects of severe malaria in endemic areas but few data are available for imported malaria. Therefore, determinants of severe imported malaria are not well known. The majority of patients hospitalized in the ICU for severe malaria are white caucasians as well as those patients who die.

The present study has two main objectives:

(i) to describe the clinical spectrum of severe imported malaria and to assess outcome (mortality and neurological sequelae), and the biological interactions between host and the parasite,

(ii) to evaluate the role of gene polymorphisms, of parasitic factors in the occurrence of severe malaria with a case control study comparing severe and non-severe malaria in patients matched according to ethnic patterns. The intensity of the inflammatory response will also be studied in the two groups of patients.

DETAILED DESCRIPTION:
Plasmodium falciparum malaria remains a major public health problem in endemic areas, with approximately 2 million deaths each year, especially in tropical African countries.

In non-endemic industrialized areas, imported malaria is generally diagnosed in travelers, as well as immigrants from endemic countries. Such imported cases have increased worldwide, with approximately 7000 cases each year in France. Among these cases, 300 are severe requiring hospitalization in ICU with an overall mortality rate of 10%, despite available effective care.

Many studies have been performed to evaluate clinical and physiopathological aspects of severe malaria in endemic areas but few data are available for imported malaria. Therefore, determinants of severe imported malaria are not well known. The majority of patients hospitalized in ICU for severe imported malaria are white caucasians, as well as those patients who die.

The present two-year prospective multicentric nationwide study has two main objectives:

1. To describe the clinical spectrum of severe imported malaria in France and to assess outcome (especially mortality, very severe cases, and neurological sequelae).
2. To analyse the biological interactions between host and the parasite, by evaluating: the role of gene polymorphisms of the host including haemoglobin analysis, the intensity of inflammatory response, endothelial activation, and finally several plasmodial factors.

We hope to include 150 to 200 patients with severe malaria hospitalized in ICU and 150 to 200 patients with uncomplicated malaria. These two groups will be included in a case control study comparing severe and non-severe malaria with matching according to ethnic patterns.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria in Severe Malaria Group:

* Hospitalization in the ICU and
* Presence of asexual forms of Plasmodium falciparum in the blood and
* One or more severe manifestations according to the World Health Organization (WHO) definition of severe falciparum malaria published in 2000

Inclusion Criteria in Uncomplicated Malaria Group:

* Hospitalization in Medicine unit or ambulatory and
* Presence of asexual forms of Plasmodium falciparum in the blood and
* Absence of any severe manifestation according to the WHO definition of severe falciparum malaria published in 2000 with the exception of the criteria hyper parasitaemia (superior4%) when isolated or the criteria jaundice /total bilirubin superior 5 micromol/L when isolated

Exclusion Criteria:

* Patient < 18 years-old
* Impossible to obtain informed consent
* Curative treatment of malaria for more than 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe malaria and patients with uncomplicated malaria
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bruneel, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Ch Versailles, Le Chesnay, France

REFERENCES:
- [Result] Bruneel F, Hocqueloux L, Alberti C, Wolff M, Chevret S, Bedos JP, Durand R, Le Bras J, Regnier B, Vachon F. The clinical spectrum of severe imported falciparum malaria in the intensive care unit: report of 188 cases in adults. Am J Respir Crit Care Med. 2003 Mar 1;167(5):684-9. doi: 10.1164/rccm.200206-631OC. Epub 2002 Oct 31. PMID 12411286